CLINICAL TRIAL: NCT02674113
Title: Use of Regional Anesthesia in Hip Arthroscopy
Brief Title: Regional Anesthesia in Hip Arthroscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: determined not to be feasible at our site
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Ajay Aggarwal, Assistant Professor of Orthopedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1211908
Record Dates: First submitted 2015-11-07; First posted 2016-02-04 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- regional anesthesia bupivacaine (Active Comparator): regional anesthesia (a single shot fascia iliaca block using bupivacaine) prior to hip arthroscopy
  Interventions: Drug: regional anesthesia bupivacaine
- regional anesthesia placebo (Placebo Comparator): subcutaneous injection procedure placebo (0.9% sodium chloride in water)
  Interventions: Drug: regional anesthesia placebo

INTERVENTIONS:
Drug: regional anesthesia bupivacaine — a single shot fascia iliaca block using bupivacaine prior to hip arthroscopy
  Other Names: Exparel; Sensorcaine; Marcaine
  Arms: regional anesthesia bupivacaine
Drug: regional anesthesia placebo — subcutaneous injection procedure using a normal saline placebo (0.9% sodium chloride in water)
  Other Names: Sodium Chloride Injection
  Arms: regional anesthesia placebo

SUMMARY:
The purpose of this research is to determine differences in outcomes in patients who receive regional anesthesia (a fascia iliaca block) versus placebo prior to undergoing hip arthroscopy with labral repair and/or debridement and osteoplasty for hip impingement.

DETAILED DESCRIPTION:
Methods: After informed consent is obtained at a routine/pre-surgical clinic visit, all patients who meet eligibility criteria will undergo randomization into one of two groups. These groups are 1) to receive regional anesthesia (a single shot fascia iliaca block using bupivacaine) prior to hip arthroscopy, or 2) undergo a subcutaneous injection procedure using a normal saline placebo (0.9% sodium chloride in water) instead of bupivacaine. Intra-operatively, both groups will receive general anesthesia and local anesthesia (lidocaine and bupivacaine in the peripheral compartment).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing primary hip arthroscopy with labral repair and osteoplasty for hip impingement
* Age 18-45 years old
* Not pregnant
* No history of neuropathic pain
* No radiographic signs of osteoarthritis of the operative hip (Tönnisgrade 1)
* Willing and able to comply with post-operative hip arthroscopy protocol
* No documented allergy to anesthetic agents
* Able to attend follow up appointments

Exclusion Criteria:

* Allergy to regional anesthetic
* Age <18 or >45 years
* Pregnant females
* History of neuropathic pain
* Radiographic signs of osteoarthritis (Tönnis grade 2)
* Unable to speak/understand English
* Currently imprisoned
* Unwilling/unable to provide consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Subject log to record number of pain pills taken by subject for 7 days | 7 days
  A log that is used by the subject to record how many oral pain medications they take for 7 days.

SECONDARY OUTCOMES:
Record of Pain Medication given in PACU | immediately post-op (while in PACU, on average 1-4 hours total)
  Record narcotic requirements in PACU
Harris Hip score | 6 weeks
  Patient reported outcome. These will be completed at the pre-operative and all post-operative clinic visits.
Visual analog pain scale | 6 weeks
  Patient reported outcome. These will be completed at the pre-operative and all post-operative clinic visits.
iHOT-12 (international hip outcome tool) | 6 weeks
  Patient reported outcome. These will be completed at the pre-operative and all post-operative clinic visits.
HOOS (hip disability and osteoarthritis outcome score) | 6 weeks
  Patient reported outcome. These will be completed at the pre-operative and all post-operative clinic visits.
Duration of time in PACU | immediately post-op, on average between 1-4 hours
Reported Falls Post-op | Time inpatient, on average 12-48 hours
Unplanned admissions and/or readmissions | 6 weeks
  number of unplanned admissions/readmission
Days until starting rehabilitation | immediately post-op, on average 24 hours - 2 weeks
Patient satisfaction | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Aggarwal, MD, Principal Investigator — University of Missouri Health System
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States